CLINICAL TRIAL: NCT06873607
Title: Evaluation of the Effectiveness of a Mobile Application Developed for Individuals With Rheumatoid Arthritis
Brief Title: Effectiveness Evaluation of a Mobile Application for Rheumatoid Arthritis
Acronym: RA-App
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Merve Akinci, Msc, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RA mobile app
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Rheumatoid Arthritis; Mobile Application
Keywords: rheumatoid arthritis; mobile application; nursing; quality of life; disease activity
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mobile app care (Experimental): Participants in this group will receive mobile application-supported care for 12 weeks, along with the recommended treatment. The content of the mobile application will include information about the disease, recommended lifestyle changes, as well as exercise and nutrition suggestions.
  Interventions: Device: mobile app
- Control (Other): These patients will not use the mobile application and will continue to receive standard treatment and care.
  Interventions: Other: Control (Standard treatment)

INTERVENTIONS:
Device: mobile app — Mobile application content: general information about rheumatoid arthritis (causes, symptoms, treatment), lifestyle changes, coping strategies for symptoms, nutrition and exercise recommendations, and daily life considerations.
  Other Names: standard treatment and care
  Arms: Mobile app care
Other: Control (Standard treatment) — Routine medical check-ups and the information provided during these visits
  Arms: Control

SUMMARY:
The aim of this experimental study is to develop a mobile application for patients with rheumatoid arthritis based on evidence-based recommendations and to evaluate the effectiveness of the developed application.

Research Questions

1. Is the mobile application developed for patients with rheumatoid arthritis effective in improving their quality of life?
2. Is the mobile application developed for patients with rheumatoid arthritis effective in reducing their disease activity? The researchers will enable the intervention group to use the mobile application in order to assess its effectiveness, while the control group will receive routine care throughout the study period.

Participants in the intervention group will use the mobile application for 12 weeks. Changes in the parameters determined by the researchers will be examined before and after the usage period. Patients in the control group will be evaluated after the initial consultation and at the end of 12 weeks. At the conclusion of the study, the control group will also be provided access to the mobile application.

DETAILED DESCRIPTION:
The mobile application will include general information about the disease, written and audio materials on disease management, as well as videos on exercise and nutrition recommendations. Stratified randomization based on disease activity will be applied to determine the patients in the intervention and control groups. Patients in the intervention group will be encouraged to use the content available in the application through pre-programmed smartphone notifications.

Data collection forms, including the Patient Sociodemographic and Medical Characteristics Form, Disease Activity Score 28 (DAS-28), The Rheumatoid Arthritis Quality of Life Questionnaire (RAQoL), Mediterranean Diet Adherence Screener (MEDAS), International Physical Activity Questionnaire Short Form (IPAQ-SF), Bristol Rheumatoid Arthritis Fatigue Multi-Dimensional Questionnaire (BRAF-MDQ-T), Perceived Stress Scale (PSS-14), Adaptation to Chronic Illness Scale (ACIS), and Visual Analog Scale (VAS) for Pain Assessment, will be administered at the initial encounter with the patients and again after 12 weeks, as specified in the methods section.

The collected data will be analyzed using the SPSS program. After the study is completed, the mobile application will be installed on the smartphones of the patients in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older
* Diagnosis of Rheumatoid Arthritis according to the American College of Rheumatology (ACR) 1987 criteria
* Receiving stable treatment for the last 3 months with no new treatments added at the last check-up
* Ability to read and write in Turkish
* Ownership of a personal smartphone with internet connectivity and the ability to use an application
* Willingness to participate in the study

Exclusion Criteria:

* Pregnancy or breastfeeding
* Having a diagnosis of inflammatory diseases or a disease that may significantly affect the functional status (such as Multiple Sclerosis, stroke, Systemic Lupus Erythematosus, Ankylosing Spondylitis, Psoriatic Arthritis)
* Not having any neurological or psychiatric disease/problem diagnosed by a physician
* Wanting to withdraw from the study
* Exiting during the study process
* Not logging in to the mobile application once a week during the study implementation period (twelve weeks) for the intervention group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease Activity Score 28 | Baseline and 12 weeks after intervention
  It is a scoring system used to determine the disease activity of rheumatoid arthritis. Calculation is made by evaluating the number of tender and swollen joints, erythrocyte sedimentation rate, global assessment of the patient, and VAS measurements using a special type of calculator. Based on the obtained DAS score, DAS 28 ≤ 2.4 is considered remission, 2.4-3.6 indicates low disease activity, 3.6-5.5 indicates moderate disease activity, and ≥ 5.5 is classified as high disease activity.
The Rheumatoid Arthritis Quality of Life Questionnaire-RAQoL | Baseline and 12 weeks after intervention.
  It will evaluate the quality of life of individuals with rheumatoid arthritis.The obtained result ranges from 0 to 30, with higher scores indicating poorer quality of life.

SECONDARY OUTCOMES:
Mediterranean Diet Adherence Screener-MEDAS | Baseline and 12 weeks after intervention
  It consists of 14 items regarding the type of essential fat individuals use in meals, daily olive oil consumption, daily fruit and vegetable portions, daily margarine/butter and red meat consumption, weekly red wine, legumes, fish-seafood, nuts, cakes, and tomato sauce with olive oil consumption. It will be used to evaluate individuals' compliance with the Mediterranean diet. After assigning 1 or 0 points to each item based on the consumption amount, the total score is calculated. A score of ≤ 5 indicates low adherence, 6-9 indicates moderate adherence, and ≥ 10 indicates high adherence.
International Physical Activity Questionnaire Short Form-IPAQ-SF | Baseline and 12 weeks after intervention
  It provides information about the time individuals spend in light, moderate, and vigorous activities and the time they spend sitting. It will be used to determine the physical activity level of individuals. For each activity level, the MET (Metabolic Equivalent) value is multiplied by the number of days and minutes, resulting in a "MET-min/week" score. The obtained value is classified as physically inactive (MET ≤ 600 energy level), insufficiently active (MET = 600-3000 energy level), and sufficiently active (MET ≥ 3000 energy level).
The Stanford Health Assessment Questionnaire-HAQ | Baseline and 12 weeks after intervention
  It is a scale that questions how rheumatological diseases affect the daily lives of individuals.A higher score on the scale indicates functional impairment. The questionnaire assesses the past week and evaluates the patient's difficulty in performing certain activities.
Bristol Rheumatoid Arthritis Fatigue Multi-Dimensional Questionnaire-BRAF-MDQ-T | Baseline and 12 weeks after intervention
  It will be used to determine the fatigue level of individuals with rheumatoid arthritis. It consists of four different subgroups: physical fatigue, fatigue in daily living activities, cognitive fatigue, and emotional fatigue.A higher score on the scale indicates increased fatigue.
Perceived Stressed Scale-PSS-14 | Baseline and 12 weeks after intervention
  It will be used to assess patients' perception of stress.A higher score indicates a greater perception of stress.
Adaptation to Chronic Illness Scale-ACIS | Baseline and 12 weeks after intervention
  This scale was developed to assess the adaptation process of individuals with chronic diseases to their illness. It evaluates factors such as patients' compliance with treatment, adaptation to lifestyle changes, and how they cope with the difficulties brought about by the disease.Higher scores on the overall scale and its subdimensions indicate a higher level of adaptation to the illness.
Visual Analog Skala-VAS | Baseline and 12 weeks after intervention
  It will be used to assess the severity of pain experienced by patients. The pain intensity assessment is typically conducted using a 10 cm (100 mm) long horizontal or vertical line, starting with "No Pain" and ending with "Unbearable Pain." The patient marks the appropriate point on the line based on their perceived pain. In this study, the responses provided by patients regarding their pain intensity will be quantified using a 100 mm scale.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - University of Health Science Gulhane Training and Research Hospital, Ankara, Yahşihan
  - University of Health Science Gulhane Training and Research Hospital, Ankara

IPD SHARING:
Plan to Share IPD: No
The sharing of individual patient data is not feasible due to the sensitive nature of the data and the potential risks of re-identification, which could compromise patient confidentiality. The study design and the intended use of the data do not require IPD sharing. The focus will be on aggregate analysis and summary results, which do not involve the release of individual patient-level data.